CLINICAL TRIAL: NCT03278899
Title: A Non-interventional Study to Prospectively Assess Baseline Status and Disease Progression in Male Children With X-Linked Adrenoleukodystrophy
Brief Title: A Study to Prospectively Assess Disease Progression in Male Children With X-ALD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: NeuroVia, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: NV1205-008
Record Dates: First submitted 2017-08-30; First posted 2017-09-12 (Actual); Last update posted 2018-08-08 (Actual); Status verified 2018-05

CONDITIONS: X-Linked Adrenoleukodystrophy
Keywords: Adrenoleukodystropy; X-ALD; ALD
MeSH Terms: conditions — Adrenoleukodystrophy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biospecimen retained: Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a non-interventional, multi-center study that follows general principles of periodic assessment of X-ALD patients in routine practice. No study drug treatment will be given and no changes to patient treatment are necessary.

DETAILED DESCRIPTION:
This is a non-interventional, multi-center study that follows general principles of periodic assessment of X-ALD patients in routine practice. No study drug treatment will be given and no changes to the patient treatment are necessary.

Patients with X-ALD will be recruited and invited to attend a baseline visit. After eligible patients are enrolled, retrospective and baseline data will be collected. After enrollment, patients will be seen approximately every 6 months until they meet withdrawal criteria or the Sponsor terminates the study.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent by patient's parent(s)/legally acceptable representative(s). In addition, signed children's assent form according to local requirements.
* Males patients 2-13 years of age with a confirmed diagnosis of X-ALD that fall into one of the following:

  * Asymptomatic patients without MRI evidence of cerebral involvement
  * Patients with MRI evidence of cerebral involvement (Loes score ≥0.5) with or without clinical symptoms
  * Patient who have HSCT within 3 months from enrollment

Exclusion Criteria:

* Patients who are 14 years of age or older
* Patients who are in a vegetative state
* Patients (or their guardians) who are unwilling or unable to comply with the study procedures
* Patients who received HSCT more than 3 months before enrollment

Ages: 2 Years to 13 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child
Gender Based: Yes — Males with a confirmed diagnosis of X-ALD with or without MRI evidence of cerebral involvement
Study Population: Patients will be selected from participating sites, referring physicians, and outreach communities
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2018-02-16 (Actual); Primary Completion 2021-06-01 (Estimated); Study Completion 2021-06-01 (Estimated)

PRIMARY OUTCOMES:
Loes score | baseline and 24 weeks
  Percent change from baseline in brain lesions assessed as Loes score will be calculated
Plasma VLCFA levels | baseline and 24 weeks
  Change from baseline plasma VLCFA levels
Neurological symptoms | baseline and 24 weeks
  Development of new neurological symptoms throughout the study

CONTACTS AND LOCATIONS:
Overall Officials: John Henderson, MD, Study Director — NeuroVia, Inc.
Locations (3):
- United States (3):
  - Stanford University, Palo Alto, California
  - Massachusetts General Hospital, Boston, Massachusetts
  - University of Pittsburgh, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No